CLINICAL TRIAL: NCT02576262
Title: HPV Integration Testing for Human Papillomavirus-Positive Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Chief Physician, Huazhong University of Science and Technology
Other Study IDs: CCS-02
Record Dates: First submitted 2015-09-22; First posted 2015-10-15 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HPV-positive women，30-65 years of age
  Interventions: Procedure: TCT，HPV，colposcopic inspection

INTERVENTIONS:
Procedure: TCT，HPV，colposcopic inspection

SUMMARY:
Papanicolaou (Pap) triage, with high specificity, has been recommended for primary Human papillomavirus (HPV) testing but is flawed by poor sensitivity and cytologist dependence. the investigators evaluated the potential role of HPV Integration detection in cervical exfoliated cells in HPV-positive women from a clinic-based population.

ELIGIBILITY:
Inclusion Criteria:

Women aged 30-65 years old visiting the gynecologic clinic of hospital

Exclusion Criteria:

1. Not providing informed consent
2. previously confirmed CIN, cervical cancer, or other malignancies
3. previous therapeutic procedure to cervix
4. pregnancy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants who visited the gynecologic clinic of hospital for various gynecologic disorders and underwent primary HPV testing were prospectively recruited
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the HPV integration screening test with comparison to HPV testing or TCT | 14 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD, PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China